CLINICAL TRIAL: NCT02961673
Title: A Phase I/Ⅱ Clinical Trial to Compare the Safety and Efficacy of HU-014 Versus Botox® in Subject With Moderate to Severe Glabellar Lines
Brief Title: The Safety and Efficacy Study of HU-014 Versus Botox® in Subject With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HU-014_P1/2
Record Dates: First submitted 2016-09-26; First posted 2016-11-11 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Glabellar Lines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HU-014 Inj(Phase 1 and 2) (Experimental): HU-014 Inj was given an injection to 5 glabellar lines each 4 U/0.1ml (Total 20 U/0.5ml, IM)
  Interventions: Biological: HU-014 Inj
- Botox Inj(Phase 2) (Active Comparator): Botox Inj was given an injection to 5 glabellar lines each 4 U/0.1ml (Total 20 U/0.5ml, IM)
  Interventions: Biological: Botox Inj

INTERVENTIONS:
Biological: HU-014 Inj — Clostridium botulinum type A
  Arms: HU-014 Inj(Phase 1 and 2)
Biological: Botox Inj — Clostridium botulinum type A
  Arms: Botox Inj(Phase 2)

SUMMARY:
A Phase I/Ⅱ Clinical Trial to Compare the Safety and Efficacy of HU-014 versus Botox® in Subject with Moderate to Severe Glabellar Lines

ELIGIBILITY:
Inclusion Criteria:

* Facial Wrinkle Scale (FWS) score > 2 when Subject knits brow extremely

Exclusion Criteria:

* Volunteer who has history of any diseases following. (myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis etc.)
* From screening, Subject who get a plastic Surgery including fascioplasty, Prosthesis implantation within 6 Weeks
* Subject who has skin disorder including infection and scar on injection site
* Subject who takes a medication including skeletal muscle relaxants, Aminoglycoside, lincomycin, anticholinergic drug, benzodiazepine, benzamide etc.
* Subject who takes a medication including anticoagulant, antithrombotic drug except low dose aspirin (below 325 mg/day)
* Any condition that, in the view of the investigator, would interfere with study participation

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Assessment of Treatment-Emergent Adverse events (TEAs), Adverse Drug Reactions (ADRs) and Serious Adverse Events (SAEs) after injecting Investigational Product(Phase 1) | Week 4
Change from Baseline of Glabellar Lines improvement rate(Frown) | Week 4

SECONDARY OUTCOMES:
Assessment of Columbia Suicide Severity Rating Scale(C-SSRS) | Week 4, Week 8, Week 12
change from Baseline of Glabellar Lines improvement rate (Frown) | Week 8, Week 12
change from Baseline of Glabellar Lines improvement rate (Not frown) | Week4, Week 8, Week 12
Efficacy Outcome Measure (Phase 2) by colleting Subject Satisfaction assessment | Week 4, Week 8, Week 12
Assessment of TEAs (Treatment-Emergent Adverse events), ADRs (Adverse Drug Reactions) and SAEs (Serious Adverse Events) after injecting Investigational Product | Week 4, Week 8, Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No